CLINICAL TRIAL: NCT01426256
Title: Vitamin D for Enhancing the Immune System in Cystic Fibrosis
Brief Title: Vitamin D for Enhancing the Immune System in Cystic Fibrosis (DISC Study)
Acronym: DISC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Principal Investigator, Vin Tangpricha, MD, PH.D, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00052829; TANGOR11A0 (Other: Other)
Record Dates: First submitted 2011-08-29; First posted 2011-08-31 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Cystic Fibrosis; Respiratory Tract Infections
Keywords: vitamin D; cholecalciferol; cystic fibrosis; respiratory tract infection; immunity; intervention studies; inflammation; dietary supplements; alpha-Defensins; Cytokines; mortality; biological markers; Biomedical Research
MeSH Terms: conditions — Cystic Fibrosis; Respiratory Tract Infections; Inflammation | interventions — Cholecalciferol; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cholecalciferol (Vitamin D3) (Experimental): Patients will be given 250,000 IU cholecalciferol in one bolus oral dose while they are in the hospital. Three months after the initial bolus dose, patients will take 50,000 IU oral cholecalciferol every other week for 9 months.
  Interventions: Dietary Supplement: Cholecalciferol
- Placebo (No Intervention): Patients will be given placebo pills in one bolus oral dose while they are in the hospital. Three months after the initial bolus dose, patients will take a placebo pill every other week for 9 months.

INTERVENTIONS:
Dietary Supplement: Cholecalciferol — Bolus dose of 250,000 IU during hospitalization + maintenance dose of 50,000 IU vitamin D every other week to be initiated 3 months after bolus dose
  Other Names: Vitamin D
  Arms: Cholecalciferol (Vitamin D3)

SUMMARY:
The purpose of this study is determine if high-dose vitamin D supplementation improves clinical outcomes related to lung function and immunity in patients with Cystic Fibrosis who are admitted to the hospital with an acute lung infection.

DETAILED DESCRIPTION:
Patients with Cystic Fibrosis (CF) have a shorter life span than the general population due to complications with lung infections, which eventually progress to lung failure. New research has suggested that high levels of vitamin D may be protective against lung infections and may promote the action of anti-bacterial proteins needed to ward off infections. Research has also suggested that high vitamin D levels are linked to lower mortality rates; however these hypotheses have not been adequately studied in patients with CF. An investigation of the effects of vitamin D supplementation is of particular interest in this population because patients with CF generally have high rates of vitamin D deficiency. The investigators have preliminary data from a previous study suggesting that vitamin D supplementation in patients with CF lowers markers of inflammation, promotes anti-bacterial proteins, and reduces mortality. In this proposed multi-center study the investigators will examine the effects of a high dose vitamin D supplementation on patients with CF who are admitted to the hospital for lung infection. The investigators will use a randomized, placebo-controlled trial design to determine if mortality and infection rates over 1 year are reduced in patients who receive the high-dose vitamin D supplementation compared to those who receive placebo. The investigators will also determine if vitamin D affects markers of inflammation and anti-bacterial proteins, as well as CF-related clinical outcomes, such as lung function. The investigators plan to recruit 280 adults and adolescents with CF (ages > 16yrs), with approximately 150 subjects recruited at Emory (Emory University Hospital and Children's Healthcare of Atlanta). Participants will initially be seen by the study researchers during the first week of in-patient hospitalization, and they will be followed over the course of one year during their regularly-scheduled out-patient CF clinic visits. The treatment group will receive an initial oral bolus dose of 250,000 IU vitamin D, and at 3 months follow-up they will receive 50,000 IU vitamin D every other week. Current CF Guidelines for vitamin D supplementation recommend a daily intake of 800 IU of vitamin D per day, therefore in addition to the vitamin D or placebo they receive at the beginning of the study and at 3 months, all participants will receive 800 IU of vitamin D daily. If our hypotheses are correct, this study has potential for reducing infection and promoting survival in patients with CF using vitamin D, a relatively inexpensive supplement.

ELIGIBILITY:
Inclusion Criteria:

* Adult and adolescent CF patients
* age >16 years
* admitted to the inpatient hospital setting for a pulmonary exacerbation of cystic fibrosis
* enrolled within 72 hours of admission
* able to tolerate oral medications
* expected to survive hospitalization

Exclusion Criteria:

* Inability to obtain or declined informed consent from the subject and/or legally authorized representative
* History of serum 25(OH)D >55 ng/mL in the past 12 months
* History of serum 25(OH)D <10 ng/mL in the past 12 months
* Current intake of more than 2,000 IU of vitamin D
* intake of 2,000 IU of vitamin D or its equivalent weekly dose (14,000 IU) for more than 1 week at any time within the past 60 days or intake of greater than vitamin D 10,000 IU once at anytime in the past 60 days
* Pregnancy or plans to become pregnant during the course of the study (12 months)
* History of disorders associated with hypercalcemia including parathyroid disease
* Current hypercalcemia (albumin-corrected serum calcium >10.8 mg/dL or ionized calcium >5.2 mg/dL)
* History of nephrolithiasis
* Chronic kidney disease worse than stage III (<60 ml/min)
* Oral or intravenous glucocorticoid use currently or in the past month
* History of lung transplantation or awaiting lung transplant
* patient in hospice care
* FEV1% predicted <20%
* Current significant hepatic dysfunction total bilirubin > 2.5 mg/dL with direct bilirubin > 1.0 mg/dL
* Current use of cytotoxic or immunosuppressive drugs
* History of AIDS
* History of illicit drug abuse (defined as history of enrollment into a drug rehabilitation program or hospital visits due to drug use within the past 3 years or any use of the following drugs in the past 6 months (cocaine, opiates, amphetamines, marijuana) or any positive toxicology screen for (cocaine, opiates, amphetamines, marijuana)
* Previous enrollment in the study
* Current enrollment in another intervention trial
* Too ill to participate in study based on investigator's or study team's opinion

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2011-10; Primary Completion 2017-04 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Study enrollment to next pulmonary exacerbation requiring any antibiotics, hospitalization or death. | 12 months

SECONDARY OUTCOMES:
inflammation | 12 months
  We will examine whether the high-dose vitamin D treatment regimen decreases the pro-inflammatory cytokines, IL-6, IL-8, and TNF- α.
mortality as a separate outcome | 12 months
re-hospitalization as a separate outcome | 12 months
anti-microbial proteins | 12 months
  We will examine whether the high-dose vitamin D treatment regimen increases cathelicidin and hBD-2 mRNA expression in both peripheral blood mononuclear cells (PBMCs) and induced sputum (by quantitative PCR).
Lung function | 12 months
  We will examine whether high dose vitamin D improves serial lung function, as measured by FEV1
Antibiotic use | 12 months
  Rates of pulmonary exacerbation requiring antibiotics due to presumed infection after 12 month
glucose metabolism | 12 months
  Rates of new onset diabetes and mean glucose values in each group

CONTACTS AND LOCATIONS:
Overall Officials: Vin Tangpricha, MD, PhD, Principal Investigator — Emory University
Locations (5):
- United States (5):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Emory Hospital, Atlanta, Georgia
  - University of Iowa, Iowa City, Iowa
  - University of Cincinnati, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio

REFERENCES:
- [Background] Wolfenden LL, Judd SE, Shah R, Sanyal R, Ziegler TR, Tangpricha V. Vitamin D and bone health in adults with cystic fibrosis. Clin Endocrinol (Oxf). 2008 Sep;69(3):374-81. doi: 10.1111/j.1365-2265.2008.03216.x. Epub 2008 Feb 11. PMID 18284636
- [Background] Khazai NB, Judd SE, Jeng L, Wolfenden LL, Stecenko A, Ziegler TR, Tangpricha V. Treatment and prevention of vitamin D insufficiency in cystic fibrosis patients: comparative efficacy of ergocalciferol, cholecalciferol, and UV light. J Clin Endocrinol Metab. 2009 Jun;94(6):2037-43. doi: 10.1210/jc.2008-2012. Epub 2009 Mar 31. PMID 19336509
- [Background] Pepper KJ, Judd SE, Nanes MS, Tangpricha V. Evaluation of vitamin D repletion regimens to correct vitamin D status in adults. Endocr Pract. 2009 Mar;15(2):95-103. doi: 10.4158/EP.15.2.95. PMID 19342361
- [Derived] Tangpricha V, Lukemire J, Chen Y, Binongo JNG, Judd SE, Michalski ES, Lee MJ, Walker S, Ziegler TR, Tirouvanziam R, Zughaier SM, Chesdachai S, Hermes WA, Chmiel JF, Grossmann RE, Gaggar A, Joseph PM, Alvarez JA. Vitamin D for the Immune System in Cystic Fibrosis (DISC): a double-blind, multicenter, randomized, placebo-controlled clinical trial. Am J Clin Nutr. 2019 Mar 1;109(3):544-553. doi: 10.1093/ajcn/nqy291. PMID 30793177